CLINICAL TRIAL: NCT05735613
Title: The Efficacy of Different Techniques of Crestal Sinus Lifting to Place Dental Implant Into Prosterior Maxilla of Deficient Height: Randomised Clinical Trial
Brief Title: Efficacy of Different Techniques of Crestal Sinus Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Halim Hashem, assistant lecturer of periodontology and oral medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410/293
Record Dates: First submitted 2022-03-18; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Maxillary Sinus Augmentation
Keywords: deficient posterior maxilla; crestal sinus lift; dental implant; bone density; bone graft; maxillary sinus augmentation

STUDY DESIGN:
Intervention Model Description: The patients divided into 3 groups:
  Group 1:7patients treated by traditional closed sinus lift (osteotome) with bone grafting (xenograft) and implant placement.
  Group 2:7patients treated by densah drills(Versah, Jackson, MI, USA) sinus lift with bone grafting (xenograft) and implant placement.
  Group 3:7patients treated by piezoelectric (Piezotome; Satelec) crestal sinus lift with bone grafting (xenograft) and implant placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Osteotome crestal sinus lifting (Experimental): Full thickness flap elevated, then elevation of sinus floor by Osteotome, then adding the bone graft and implant placement. Measuring the ISQ value by Ostell device then flap sutured. After 6 months of implant placement exposure of implant for prosthetic phase and measuring secondary stability.
  Interventions: Procedure: osteotome crestal sinus lifting
- osseodensification crestal sinus lifting (Experimental): Full thickness flap elevated, then elevation of sinus floor by Densah burs, then adding the bone graft and implant placement. Measuring the ISQ value by Ostell device then flap sutured. After 6 months of implant placement exposure of implant for prosthetic phase and measuring secondary stability.
  Interventions: Procedure: osseodensification crestal sinus lifting
- peizoelectric crestal sinus lifting (Experimental): Full thickness flap elevated, then elevation of sinus floor through piezoelectric surgery via intralift kit, then adding the bone graft and implant placement. Measuring the ISQ value by Ostell device, followed by flap suturing. After 6 months of implant placement exposure of implant for prosthetic phase and measuring secondary stability.
  Interventions: Procedure: piezoelectric crestal sinus lifting

INTERVENTIONS:
Procedure: osteotome crestal sinus lifting — Full thickness flap elevated to expose the crest of alveolar ridge. Pilot drill used to start the osteotomy preparation, which should be ended 1mm short of sinus floor. The drills can be sequentially used to widen the osteotomy site to the same level (1 mm short of the sinus floor), an osteotome of diameter a little less than the planned implant body, will be inserted in the prepared osteotomy site and gently tapped to reach the same level, the osteotome will be tapped gently to fracture up the sinus floor.Clinical check for membrane still intact, blocking the patient's nostrils and asking the patient to blow through his or her nose. Xenograft will be added as the grafting material and pushed to the sinus through the osteotomy site until the desired height of sinus elevation will be gained, the implant fixture will be inserted. Smart peg will be placed on implant and Ostell will be used to record ISQ.
  Arms: Osteotome crestal sinus lifting
Procedure: osseodensification crestal sinus lifting — Full thickness flap elevated to expose the crest of alveolar ridge. Pilot drill used to start the osteotomy preparation, which should be ended 1mm short of sinus floor. Change the drill motor to reverse-densifying Mode (counterclockwise drill speed 800-1500 rpm with copious irrigation), Begin with the densah bur (2.5mm) until 1 mm short of the sinus floor, use the next wider Densah Bur (3.0mm) in the same mode and advance it into the previously created osteotomy with modulating pressure and a pumping motion. When feeling the haptic feedback of the drill reaching the dense sinus floor, modulate pressure with a gentle pumping motion to advance past the sinus floor in 1 mm increments, the next wider densah drills advance in the osteotomy.Clinical check for membrane still intact. Xenograft added and pushed to the sinus through the osteotomy site then the implant fixture will be inserted.
  Arms: osseodensification crestal sinus lifting
Procedure: piezoelectric crestal sinus lifting — initial osteotomy will be performed with a 2-mm twist drill to remove the cortical bone, then the intralift tips (Intralift; TKW1, TKW2, TKW3,TKW4, TKW5; Satelec). TKW1 to TKW4 tips have diameters of 1.35 mm, 2.1 mm, 2.35 mm, and 2.8 mm and will be used to gradually widen the access canal to the Schneider membrane, gentle pressure will be applied on the tips to deepen the pathway, and a sterile spray (80 mL/min) cooling the tips to avoid heat injury. The TKW5 tip will be then inserted into the access canal, and the ultrasonic activation for 5 seconds with internal irrigation of 40 mL/min and repeated at 50 mL/min and then 60 mL/min. The sinus membrane will be pushed upward by the hydraulic pressure, the floating of the sinus membrane will be evaluated, and then the TKW4 (Ø 2.8 mm) will be used again to widen the access canal to the sinus membrane before plugging the bone graft.xenograft added. Implant fixture inserted and flap statured
  Arms: peizoelectric crestal sinus lifting

SUMMARY:
Twenty one patients with deficient posterior maxilla and alveolar bone height ≤ 5mm were included.Those patients randomly divided into 3 equal groups:

1. Group 1: 7 patients treated by osteotome closed sinus lift with bone grafting (xenograft) and implant placement.
2. Group 2: 7 patients treated by densah burs(Versah, Jackson, MI, USA) sinus lift with bone grafting (xenograft) and implant placement.
3. Group 3: 7 patients treated by piezoelectric (Piezotome; Satelec) crestal sinus lift with bone grafting (xenograft) and implant placement.

DETAILED DESCRIPTION:
Patients have been asked asked to use 0.12% chlorhexidine digluconate rinse, and Povidone iodine solution will be used to perform extraoral antisepsis. After administration of local anesthesia at the implant site, a full thickness flap was elevated to expose the crest of alveolar ridge. A pilot drill will be used to start the osteotomy preparation, which should be ended 1mm short of sinus floor.

In group 1; (closed sinus lifting with Osteotome): The drills can be sequentially used to widen the osteotomy site to the same level (1 mm short of the sinus floor), an osteotome of diameter a little less than the planned implant body, will be inserted in the prepared osteotomy site and gently tapped to reach the same level, the osteotome will be tapped gently to fracture up the sinus floor.

In group 2; (closed sinus lifting with densah drills): Change the drill motor to reverse-densifying Mode (counterclockwise drill speed 800-1500 rpm with copious irrigation), Begin with the densah bur (2.5mm) until 1 mm short of the sinus floor, use the next wider Densah Bur (3.0mm) in the same mode and advance it into the previously created osteotomy with modulating pressure and a pumping motion. When feeling the haptic feedback of the drill reaching the dense sinus floor, modulate pressure with a gentle pumping motion to advance past the sinus floor in 1 mm increments, the next wider densah drills advance in the osteotomy.

In group 3: The initial osteotomy will be performed with a 2-mm twist drill to remove the cortical bone, then the intralift tips (Intralift; TKW1, TKW2, TKW3, TKW4, TKW5; Satelec). TKW1 to TKW4 tips have diameters of 1.35 mm, 2.1 mm, 2.35 mm, and 2.8 mm and will be used to gradually widen the access canal to the Schneider membrane, gentle pressure will be applied on the tips to deepen the pathway, and a sterile spray (80 mL/min) cooling the tips to avoid heat injury. The TKW5 tip will be then inserted into the access canal, and the ultrasonic activation for 5 seconds with internal irrigation of 40 mL/min and repeated at 50 mL/min and then 60 mL/min. The sinus membrane will be pushed upward by the hydraulic pressure, the floating of the sinus membrane will be evaluated, and then the TKW4 (Ø 2.8 mm) will be used again to widen the access canal to the sinus membrane before plugging the bone graft.

For all groups: Clinical check for membrane still intact, blocking the patient's nostrils and asking the patient to blow through his or her nose. Xenograft was added as the grafting material and pushed to the sinus through the osteotomy site until the desired height of sinus elevation will be gained, the implant fixture will be inserted. Smart peg will be placed on implant and Ostell will be used to record ISQ. Cover screw will be placed on implant and flab will be sutured. Sutures were removed after 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Young and adult patients of both sexes.
2. Patients exhibit class C residual bone height according to ABC sinus augmentation classification.(18)
3. The edentulous ridges are covered with mucoperiosteum free from signs of inflammation, ulceration or scar tissue.
4. Remaining natural teeth have good periodontal tissue support.
5. Occlusion showing sufficient inter-arch and intra-arch spaces for future prosthesis.

Exclusion Criteria:

1. Patients with systemic conditions that could influence the outcome of the therapy as: Pregnancy and Heavy smokers
2. Patients with systemic disease that may affect bone quality.
3. Uncooperative patients
4. Patients with active periodontal disease.
5. Patients with neglected oral hygiene.
6. Patients with limited mouth opening and unfavorable intermaxillary arch space.
7. Patients with maxillary sinus disease or previous sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
dental implant stability | 6 months
  evaluation of implant primary and secondary stability clinically using ostell device through measuring ISQ value
maxillary sinus augmentation | 6 months
  evaluation of vertical bone gain using CBCT before and after six months of implant placement

SECONDARY OUTCOMES:
bone density | 6 months
  measuring bone density before and after 6 months of implant placement
crestal bone loss | 6 months
  crestal bone loss after 6 months of implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H. Hashem, Ass.Leturer, Principal Investigator — Al-Azhar University
Locations (1):
- The Faculty of Dentistry- AL-AZHAR University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vercellotti T, De Paoli S, Nevins M. The piezoelectric bony window osteotomy and sinus membrane elevation: introduction of a new technique for simplification of the sinus augmentation procedure. Int J Periodontics Restorative Dent. 2001 Dec;21(6):561-7. PMID 11794567
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Result] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT05735613/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT05735613/SAP_001.pdf